CLINICAL TRIAL: NCT01765218
Title: Topiramate as an Adjuvant to Therapeutic Hypothermia for Infants With Hypoxic Ischemic Encephalopathy
Brief Title: Topiramate in Neonates Receiving Whole Body Cooling for Hypoxic Ischemic Encephalopathy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped early due to changes in the UC Davis guidelines on who qualified for therapeutic hypothermia and significant difficulty in recruitment of patients following the COVID19 pandemic.
Sponsor: Kristin R Hoffman (Other)
Responsible Party: Sponsor-Investigator, Kristin R Hoffman, Assistant Professor of Clinical Pediatrics, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1182678
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic ischemic encephalopathy; HIE; Perinatal depression; Whole body cooling; Therapeutic hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive the standard of care intervention for HIE at our institution (whole body cooling for 72h followed by gradual rewarming)
  Interventions: Drug: Placebo
- Topiramate (Active Comparator): In addition to whole body cooling, infants assigned to the topiramate group will receive 5mg/kg of topiramate daily enterally for a total of 5 doses. The first dose will be administered as soon as possible on admission.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Infants assigned to the topiramate group will receive 5mg/kg of topiramate daily enterally for a total of 5 doses. The first dose will be administered as soon as possible on admission.
  Other Names: Topamax; Topiragen
  Arms: Topiramate
Drug: Placebo — A placebo identical in appearance to the active agent (topiramate)
  Arms: Placebo

SUMMARY:
The goal is to see whether topiramate (an anti-epileptic agent) improves the outcome of babies with neonatal hypoxic encephalopathy who are receiving whole body cooling.

DETAILED DESCRIPTION:
Hypoxic ischemic encephalopathy (HIE) is a devastating and unexpected disease in newborns that affects 1.5-2.6 per 1000 live births. Hypoxic ischemic encephalopathy has a mortality rate of up to 30% and survivors are at significant risk for adverse long-term outcomes, including seizures, cerebral palsy, and developmental delay. The investigators propose a randomized controlled study comparing therapeutic hypothermia alone, or therapeutic hypothermia combined with topiramate. The investigators hypothesize that adjuvant therapy with topiramate will reduce short term severity of HIE including seizures (the primary outcome), a composite HIE severity score, and reduce the time of normalization of the amplitude integrated EEG (aEEG). The investigators further hypothesize, that it will improve longer term outcomes such as developmental outcome. The primary hypothesis is that seizures before hospital discharge (or before 4 weeks post-natal age (which ever is earlier)) will be significantly reduced in the topiramate group compared to the control group

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for cooling the baby must meet all three of the following sets of criteria

1. Be near term (typically ≥34wks gestation) and be aged < 6h old
2. Have signs of early perinatal depression (EITHER 10 minute Apgar score < 5, OR pH < 7.00 within 60mins of age, OR Base Excess < -12 within 60mins of age, OR need respiratory support at 10min of age due to respiratory depression)
3. Have signs of moderate or severe encephalopathy based on either clinical examination or on amplitude integrated aEEG assessment

Exclusion Criteria:

1. Known congenital myopathy
2. Known congenital neuropathy

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin R Hoffman, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Topiramate
Started (Enrolled) | 17 | 17
Completed (Received 5 doses of Topiramate) | 16 | 15
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Topiramate | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Customized [Mean (Full Range); unit: Weeks]
  Gestational Age | 39.12 [37 to 40.71] | 38.88 [36.14 to 41.29] | 39 [36.14 to 41.29]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomization did not account for gender
  Participants
    Female | 10 | 5 | 15
    Male | 7 | 12 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Many participants marked "Other"
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 0 | 0 | 0
    White | 5 | 5 | 10
    More than one race | 3 | 1 | 4
    Unknown or Not Reported | 6 | 8 | 14
Birth Weight (g) [Mean (Full Range); unit: grams] — Birth Weight in grams Population: Birth Weight as measured in Grams between the two arms
  grams | 3236.14 [2100 to 4580] | 3159.24 [2200 to 5520] | 3197.46 [2100 to 5520]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Seizures
Description: Clinical or electrical seizures occuring before hospital discharge or before 4w post-natal age (which ever is earlier) will be compared between the topiramate and control groups.
Time Frame: At 4 weeks post-natal age or the time of hospital discharge (whichever is earlier)
Measure: Number; unit: Participants with Seizures
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 17 | 17
Participants with Seizures | 3 | 1

ADVERSE EVENTS:
Time Frame: Data was collected until discharge, typically less than one month
Description: Charts were reviewed to collect adverse event data.
Arm/Group | Placebo | Topiramate
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Topiramate (N=17)
Necrotizing Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) — Infection and necrosis of the bowel
Chronic Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Chronic Lung Disease or Bronchopulmonary Dysplasia
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Topiramate (N=17)
Need for Bronchodilator Therapy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (10) — Need for Bronchodilator Therapy (albuterol)
Need for Bicarbonate or THAM for acidosis (General disorders) | 2 (3) | 3 (6) — Need for Bicarbonate or THAM for acidosis

LIMITATIONS AND CAVEATS:
Study was stopped short of intended recruitment due to difficulty with recruitment during COVID pandemic and changes to the therapeutic hypothermia protocol at our institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT01765218/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT01765218/ICF_001.pdf